CLINICAL TRIAL: NCT06773221
Title: A Key Therapeutic System for Reversing MAFLD-related Cirrhosis: a Randomized Double-blind Controlled Trial on the Efficacy and Safety of Chiglitazar in Patients with MAFLD-related Cirrhosis
Brief Title: The Efficacy and Safety of Chiglitazar in Patients with MAFLD-related Cirrhosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Friendship Hospital (Other)
Collaborators: Beijing Ditan Hospital (Other); Peking University People's Hospital (Other); Beijing YouAn Hospital (Other)
Responsible Party: Principal Investigator, Hong You, Vice president of hospital, Beijing Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-P2-487-01
Record Dates: First submitted 2025-01-02; First posted 2025-01-14 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Metabolic Dysfunction Associated Fatty Liver Disease; Compensated Liver Cirrhosis
MeSH Terms: interventions — chiglitazar

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment arm (Experimental): Chiglitazar 64mg, oral, qd, for 72 weeks
  Interventions: Drug: Chiglitazar 64mg
- Control arm (Placebo Comparator): Placebo, oral, qd, for 72 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Chiglitazar 64mg — Chiglitazar 64mg, oral, qd, for 72 weeks
  Arms: Treatment arm
Drug: Placebo — Placebo, oral, qd, for 72 weeks
  Arms: Control arm

SUMMARY:
A total of 195 adult patients with biopsy-proven or clinically diagnosed metabolic dysfunction-associated with fatty liver disease(MAFLD)-related cirrhosis will be randomly divided into two arms. One arm will receive Chiglitazar(64 mg) treatment, while the other arm will receive placebo treatment, lasting for 72 weeks. Both the researchers and the participants will be blinded. The primary outcome is the reversal rate of cirrhosis assessed by magnetic resonance elastography. Secondary outcomes include outcome events, changes in histopathological fibrosis stage, non-invasive fibrosis tests, glucose and lipid metabolism indicators.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged between 18 and 75 years (inclusive) who understand and sign informed consent forms; 2. Compensated MAFLD-related cirrhosis diagnosis(meet one of the following conditions):

1. The liver biopsy during the screening period (liver biopsy within 6 months of screening is acceptable) showing cirrhosis with steatohepatitis according to the Non Alcoholic Fatty Liver Disease Clinical Research Network (NASH-CRN) scoring system, and there is no evidence of competitive aetiology.
2. The liver biopsy during the screening period (liver biopsy within 6 months of screening is acceptable) showing cirrhosis with steatosis (no steatohepatitis) according to NASH-CRN scoring system, and there is no evidence of competitive aetiology. There are at least 2 coexisting metabolic comorbidities or history of metabolic comorbidities, including obesity and/or type 2 diabetes mellitus (T2DM).
3. Historical biopsy showed steatohepatitis, and now diagnosed with cirrhosis through non-invasive tests or clinical criteria (see criterion (5)-1)). There is no evidence of competing aetiology. There is at least 1 coexisting or history of metabolic comorbidity.
4. Historical biopsy showed steatosis (no steatohepatitis), and now diagnosed with cirrhosis through non-invasive tests or clinical criteria (see criterion (5)-1)). There is no evidence of competing aetiology. There are at least 2 coexisting metabolic comorbidities or history of metabolic comorbidities, including obesity and/or T2DM.
5. In the absence of biopsy, MAFLD-related cirrhosis is defined based on the following criterias:

   a. Cirrhosis is defined based on one of the following non-invasive tests(NITS): i: MRE ≥ 5kPa or VCTE-LSM ≥ 20kPa (when the patients with BMI ≥ 28kg/m2 , MRE ≥ 5kPa must also be met); ii:VCTE ≥15 kPa and <20 kPa and 1 of the following: MRE≥4.45kPa or Agile4≥0.565 or Platelets≤150,000/µL; iii: VCTE <15 kPa and 2 of the following: MRE≥4.45kPa or Agile4≥0.565 or Platelets≤150,000/µL; b. Current or previous imaging examinations have diagnosed fatty liver or controlled attenuation parameter (CAP)>288dB/m or magnetic resonance imaging proton density fat fraction (MRI-PDFF)>5%.

   c. There is no evidence of competing aetiology; d. There are at least 2 coexisting metabolic comorbidities or history of metabolic comorbidities, including obesity and/or T2DM.
6. If a participant's MAFLD-related cirrhosis diagnosis for eligibility is based on the biopsy screening period , no weight loss of ≥10% should have occurred in the same time period (based on medical history).

Exclusion Criteria:

1. Other chronic liver diseases (including but not limited to viral hepatitis, alcoholic liver disease, drug-induced liver injury, autoimmune liver disease, Wilson's disease, hemochromatosis, etc.)
2. There has been a continuous history of heavy drinking for 3 months or more current or rencent 5 years (heavy drinking is defined as >20 g/day in women and >30 g/day in men); Or researchers can not reliably quantify alcohol consumption.
3. Hepatic decompensation events (including ascites, esophageal and gastric variceal bleeding, hepatic encephalopathy, hepatorenal syndrome, spontaneous bacterial peritonitis, etc.) or hepatocellular carcinomaor.
4. History of malignant tumors within 5 years (excluding local squamous cell carcinoma of the skin or treated cervical intraepithelial neoplasia)；
5. Combination of autoimmune diseases (including but not limited to systemic lupus erythematosus, multiple sclerosis, Hashimoto's thyroiditis, etc.)；
6. Combined with severe esophageal and gastric varices and/or positive red sign accessed by endoscope；
7. History of liver transplantation or bone marrow transplantationor or listed for liver transplantation;
8. Previous (<5 years before screening)or planned (during the trial period) treatment for obesity with surgery;
9. Have obesity induced by other endocrinologic disorders (i.e. Cushing Syndrome) genetic diseases;
10. Secondary factors that can cause liver steatosis, such as malnutrition, medication, genetic metabolic diseases, etc.
11. Individuals with the following abnormal indicators:

    1. Alanine aminotransferase (ALT)>5 * ULN;
    2. Aspartate aminotransferase (AST)>5 * ULN
    3. Direct bilirubin (DBIL)>1.5 * ULN
    4. Estimated glomerular filtration rate (eGFR)<60 mL/min/1.73m2
    5. Glycated hemoglobin (HbA1c)>10%
    6. MELD score ≥ 12 or Child Pugh score ≥ 8 caused by liver disease
12. History of any type of diabetes than T2DM;
13. Participants receive more than 1 month of treatment with any of the following drugs within 6 months before screening: thiazolidinedione (TZD), glucagon like peptide-1 (GLP-1) receptor agonists, bate lipid-lowing drugs, liver selective thyroxine receptor beta (TSH - β) agonists, obeticolic acid, insulin, berberine, weight-loss drugs, amiodarone, methotrexate, systemic glucocorticoids at >5 mg/day of prednisone equivalent, tamoxifen, oestrogens at doses higher than those used for hormone replacement or contraception, anabolic steroids except testosterone replacement, valproic acid, and known hepatotoxins;
14. Participants receive the following medications unless they have received a stable dose of at least 1 month prior to screening: beta blockers, thiazide diuretics, statins, niacin, ezetimibe, thyroid hormones, metformin, dipeptidyl peptidase-4 (DPP-4) inhibitors, sodium glucose cotransporter (SGLT-2) inhibitors, sulfonylureas, gliptides, alpha glucosidase inhibitors;
15. Participating in clinical trials of other drugs or medical devices within the past 3 months.
16. Participants who demonstrate recent evidence (within 6 months prior to screening) of acute or unstable cardiovascular and cerebrovascular events events (such as hospitalisation for myocardial infarction, stroke, chronic heart failure grade IV (NYHA classification), severe arrhythmia, left ventricular hypertrophy, transient ischemic attack, and/or acute peripheral vascular events);
17. QTc (Fridericia) mean interval that is greater than 500 ms at screening (triplicate electrocardiogram [ECG]) or personal or family history of long QT syndrome;
18. Have a history of major surgery or fracture in the past 3 months;
19. Severe osteoporosis or other known bone diseases, or other conditions that may lead to fractures accessed by researchers;
20. History of lower limb or systemic edema;
21. Contraindications for MRI scans, including but not limited to: cerebral aneurysm clips, implanted nerve stimulators, implanted pacemakers or defibrillators, or the presence of artificial heart valves, cochlear implants, potentially ferromagnetic intraocular foreign bodies (such as metal shavings), other implantable medical devices (such as insulin pumps), metal shrapnel or bullets remaining in the body, severe claustrophobia, tattoos (determined by the researcher and radiologist), weight exceeding the carrying capacity of the MRI scanner, etc.;
22. Positive for human immunodeficiency virus (HIV) infection;
23. History of drug use or abuse of drugs within the 12 months prior to screening.
24. patients who have smoked heavily within the past year, with a daily intake of ≥ 30 cigarettes;
25. Pregnant or lactating women, and the woman of childbearing age who are unable or unwilling to use adequate contraception;
26. Researchers believe that patients who are not suitable to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Estimated)
Dates: Start 2025-02-05 (Estimated); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Fibrosis regression rate | 72 weeks
  20% decline in magnetic resonance elastography(MRE)

SECONDARY OUTCOMES:
Cumulative incidence of outcomes events | 72 weeks
  Cumulative incidence of outcomes events(including liver decompensation, hepatocellular carcinoma, liver transplantation, and death)
Percentage of participants acheving decline in fibrosis stage in histopathology | 72 weeks
  changes in fibrosis stage in histopathology
Number of patients with decreased scores of non-invasive liver fibrosis tests | weeks 2, 4, 8, 12, 18, 24, 32, 40, 48, and 72.
  Dynamic change of non-invasive liver fibrosis tests(including APRI、FIB-4、FAST、NFS)
Number of patients with decrease of MRE | weeks 48, and 72.
  absolute change of MRE, and percentage of patients achieving 15% decline in MRE
Number of patients with change in magnetic resonance imaging-derived proton density fat fraction(MRI-PDFF)) | weeks 48, and 72.
  absolute change in MRI-PDFF, and percentage of patients achieving 30% decline in MRI-PDFF
Number of patients with decrease of liver stiffness measurement (LSM) via vibration-controlled transient elastography (VCTE) | weeks12, 24, 48, and 72.
  Absolute change in LSM, CAP, and SSM, and percentage of patients achieving 30% decline in LSM
Number of patients with change in spleen stiffness measurement (SSM)) via vibration-controlled transient elastography (VCTE) | weeks12, 24, 48, and 72.
Number of patients with change in controlled attenuation parameter(CAP) via vibration-controlled transient elastography (VCTE) | weeks12, 24, 48, and 72.
Number of patients with decrease in glycosylated hemoglobin A1c (HbA1c) | weeks12, 24, 48, and 72.
Number of patients with change in lipidmetabolism indicators. | weeks 2, 4, 8, 12, 18, 24, 32, 40, 48, and 72.
  Dynamic changes in lipidmetabolism indicators (including triglycerides, total cholesterol, high-density lipoprotein (HDL) cholesterol, low-density lipoprotein (LDL) cholesterol, and apolipoprotein B (Apo B))
Number of patients with change of liver function indictors | weeks 2, 4, 8, 12, 18, 24, 32, 40, 48, and 72.
  Dynamic change of liver function indicators (including ALT and AST)
Number of patients with change in fast plasma glucose | weeks 2, 4, 8, 12, 18, 24, 32, 40, 48, and 72.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Beijing Ditan Hospital, Capital Medical University, Beijing, China
  - Peking University People's Hospital, Beijing, China
  - Beijing Friendship Hospital, Capital Medical University, Beijing, China
  - Beijing Youan Hospital, Capital Medical University, Beijing, China